CLINICAL TRIAL: NCT00891358
Title: A Secondary Prevention Empowerment Intervention for Young Women Living With HIV
Brief Title: Empowerment Intervention for Young Women - Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ATN 073
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-07

CONDITIONS: HIV; Empowerment; HIV Infections
Keywords: Adolescent Medicine Trials Network for HIV/AIDS Interventions; Human Immunodeficiency Virus; HIV seronegativity
MeSH Terms: conditions — Empowerment; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Focus Group (Experimental): Participants in focus groups will meet and discuss their intervention needs.
  Interventions: Behavioral: Prevention Empowerment Intervention for Young Women

INTERVENTIONS:
Behavioral: Prevention Empowerment Intervention for Young Women — Using three intervention sites, focus groups will guide the development of the intervention's framework and content areas. An initial list of content areas and potential activities for presentation to the focus groups will be developed by the protocol team by reviewing existing HIV prevention interventions that have been implemented with adolescents and young adults, as well as interventions that have targeted HIV+ populations.
  The three focus groups will be convened (1 per selected ATN site) with young women living with HIV to solicit information on their intervention needs.

SUMMARY:
This study will begin to develop a culturally appropriate secondary prevention intervention for young HIV+ women through focus groups.

Using three intervention sites, focus groups will guide the development of the intervention's framework and content areas. An intervention will be developed/adapted through the data collected in the focus groups and review of relevant interventions. The intervention aims to address the following concerns: 1) reducing the risk of young women infected with HIV transmitting the virus to their sexual partners, and 2) preventing young women infected with HIV from re-infection with a new viral strain or co-infection with another sexually transmitted disease.

DETAILED DESCRIPTION:
This study will develop/adapt a culturally appropriate secondary prevention intervention for young HIV+ women through focus groups. Using three intervention sites, focus groups will guide the development of the intervention's framework and content areas. An initial list of content areas and potential activities for presentation to the focus groups will be developed by the protocol team by reviewing existing HIV prevention interventions that have been implemented with adolescents and young adults, as well as interventions that have targeted HIV+ populations.

Three focus groups will be convened (1 per selected ATN site) with young women living with HIV to solicit information on their intervention needs. All focus groups will be digitally recorded and transcribed. Executive summaries of the groups will focus on the major themes elicited by probes that explore the proposed content and structure of the interventions. The summaries will be generated by members of the Protocol Team and based on a review and integration of data from a) focus group flip charts; b) digitally recorded comments from participants; c) digitally recorded oral summaries by moderators offered during the focus groups; and d) thematic notes taken by the assistant moderator during the focus groups. Based on the outcome of the focus groups, intervention modules will be developed and modified in collaboration with the Youth Advisory Team.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth and currently female;
* Receives services at one of the selected ATN sites or their community partners;
* HIV-infected as documented by medical record review or verbal verification with referring professional;
* Between the ages of 16-24 (inclusive) at the time of informed consent/assent;
* Ability to understand both written and spoken English; and
* Gives informed consent/assent for study participation.

Exclusion Criteria:

* Presence of active, serious psychiatric symptoms (hallucinations, thought disorder) that would impair a participant's ability to meet the study requirements;
* Visibly distraught (suicidal, homicidal, exhibiting violent behavior);
* If other serious conditions are present during screening, the Protocol Team must be consulted to determine whether enrollment may interfere with the evaluation of the protocol objectives and for permission to proceed with the enrollment; or
* Intoxicated or under the influence of alcohol or other substances at the time of study enrollment*.

  * Participants cannot be visibly under the influence at the time of consent, enrollment, or during the focus group. Intoxication at the time of the focus group will exclude participation.

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Use of focus groups for development/adaptation of a secondary prevention empowerment intervention to reduce sexual risk behavior among young women living with HIV. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — John Stroger Hospital of Cook County; Adolescent Trials Network
Locations (3):
- United States (3):
  - USF College of Medicine, Tampa, Florida
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - University of Maryland Medical School, Baltimore, Maryland

REFERENCES:
- See also: ATN Website — https://www.atnonline.org